CLINICAL TRIAL: NCT02558816
Title: A Phase I/II Trial of Obinutuzumab, ABT-199 (GDC-0199) Plus Ibrutinib in Relapsed / Refractory Mantle Cell Lymphoma Patients
Brief Title: A Trial of Obinutuzumab,GDC-0199 Plus Ibrutinib in Relapsed/Refractory Mantle Cell Lymphoma Patients
Acronym: OAsIs
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Janssen, LP (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC14_0048; 2014-003740-13 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-24 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Ibrutinib - GA101 - GDC_0199 (Experimental): STEP A:C1:Ibrutinib 560mg D2-28;GA101 1000mg day 1/2,8,15;C2-6:Ibrutinib 560mg D 1-28;GA101 1000mg D1 / C7 (Maintenance phase)-C24:Ibrutinib 560mg D1-28 (until progression);GA101 1000mg D1 every 2cycles (from C8) STEP B:C1:Ibrutinib 560mg D2-28;GA101 1000mg D1/2,8,15 / C1bis : Ibrutinib 560mg day 1-28 ; GA101 1000mg D 1 ; GDC-0199 20mg/d at W1, 50mg/d at W2, 100mg at W3, 200 mg/d at W4 / C2-6:Ibrutinib 560mg D1-28;GA101 1000mg D1;GDC-0199:400mg/d W1 and 400, 600 or 800mg/d W2-3-4 + 400, 600 or 800 mg/d C3-C6 (patients 1-12).Patients 13-24:GDC-199 400mg/d / C7(Maintenance phase)-C23:Ibrutinib 560mg D1-28 (until progression);GA101 1000mg D1 every 2 cycles (from C8);GDC:400, 600 or 800 mg D1-28 (patient 1-12).Patients 13-24 : 400mg/d STEP C:C1-C1bis=Step B; C2-6:Ibrutinib 560mg D1-28;GA101 1000mg D1;GDC:400mg/d C7 (Maintenance phase)-C23 : Ibrutinib 560mg D1-28 (-->progression);GA101 1000mg D1/2 cycles (from C8);GDC-0199 400mg/d
  Interventions: Drug: Ibrutinib + GA101 +GDC-0199

INTERVENTIONS:
Drug: Ibrutinib + GA101 +GDC-0199 — Step A : 9 patients receive the combination of Ibrutinib + GA101 Step B : 24 patients receive the combination of Ibrutinib + GA101 + GDC-0199 Step C : 15 untreated patients receive the combination of Ibrutinib + GA101 + GDC-0199
  Other Names: GA101 : Obinutuzumab; Ibrutinib; GDC-0199

SUMMARY:
This is an open label, multicenter, fixed dose and dose escalation, phase I/II study.

The study will be conducted in 3 steps. The first one (step A) will be to ensure the safety of the combination of Obinutuzumab (GA101) and Ibrutinib at fixed doses in patients with relapsed or refractory Mantle Cell Lymphoma (MCL).

A total of 9 patients have been included in the first step with grouped inclusions of three patients (safety evaluation performed at each inclusion of 3 patients).

No unacceptable toxicity has been observed during step A, thefore the second step (step B) was initiated. The aim of the second step was to determine the MTD of the GDC-0199 (400-600-800mg/d) in combination of GA101 and Ibrutinib (both respecting the previous doses) by using a Continual Reassessment Method. This dose escalation method was used until the 12th patient (3 patients included at 400mg/d of GDC-0199-(no DLT), 3 at 600mg/d- (no DLT) and 6 at 800mg/d, (not DLT reported so far). Once the last patient of the 800mg cohort is evaluated for DLT, all other patients will be treated at the dose of 400mg/d of GDC-0199.

The third step (step C) for untreated patients will be conducted at the dose of 400mg/d of GDC-0199. The aim of step C is to confirm the safety profile of the GA101 + Ibrutininb + GDC-199 combination according to step B result. 15 patients will be included in this step.

DETAILED DESCRIPTION:
The study will be conducted into 3 steps for respecting the optimal safety of the OASIS trial:

Step A :

The primary objective of step A is to evaluate the safety of the combination of GA101 + Ibrutinib at fixed doses (560 mg per day of Ibrutinib + 1000 mg of GA101), in patients with relapsed or refractory Mantle Cell Lymphoma (MCL).

Secondary objectives:

* To describe the efficacy of the combination of GA101 and Ibrutinib in terms of clinical benefits response (overall response rate, complete response rate, partial response rate Cheson 99 and 07 criteria and Working Group Revised Response Criteria for Malignant Lymphomas 14), overall survival, progression free survival.
* To describe the safety and tolerability of the combination of GA101 and Ibrutinib
* To establish a bio-bank to explore biomarkers and mechanisms of action including resistance

Step B : Step B started because no unacceptable toxicity occurred in patients included in the step A.

The primary objective of this step is to determine the maximal tolerated dose (MTD) of the GDC-0199 in addition to the GA101 and Ibrutinib in relapsed refractory MCL patients by using a Continual Reassessment Method (CRM), used up to the 12th enrolled patients. No DLT occured for the first 12 patients. Based on the most recent publications, the dose of 400mg/d will be used from the 13th to the 24th patients (no CRM used).

Secondary objectives:

* To describe the efficacy of the combination GA101, Ibrutinib and GDC-0199 in terms of clinical benefits response (overall response rate, complete response rate, partial response rate Cheson 99 and 07 criteria and Working Group Revised Response Criteria for Malignant Lymphomas 14), overall survival, progression-free survival.
* To describe the safety and tolerability of the novel combination of GDC-0199, GA101 and Ibrutinib
* To establish a bio-bank to explore biomarkers and mechanism of action including resistance

Step C :

This step has started because no unacceptable toxicity was observed during the second step.

The primary objective of this step is to confirm the safety of the combination of GA101 + Ibrutinib + GDC-199 at fixed doses (560 mg per day of Ibrutinib + 1000 mg of GA101, 400mg/d of GDC-199 ), in patients with untreated Mantle Cell Lymphoma (MCL), at end of Cycle 2.

Secondary objectives :

* To describe the efficacy of the combination GA101, Ibrutinib and GDC-0199 in terms of clinical benefits response (overall response rate, complete response rate, partial response rate cheson 99 and 07 criteria and Working Group Revised Response Criteria for Malignant Lymphomas 14), overall survival, progression-free survival.
* To describe the safety and tolerability of the novel combination of GDC-0199, GA101 and Ibrutinib
* To establish a bio-bank to explore biomarkers and mechanism of action including resistance

ELIGIBILITY:
Inclusion criteria :

* Age ≥18 for French patients and Age ≥16 for UK patients
* Step A + B : Relapsed / refractory MCL after at least one line of treatment. The relapse diagnosis (within 3 months before baseline), needs to be histologically confirmed (tumor biopsy or bone marrow biopsy) or confirmed by the presence (immunuphenotype) of circulating tumor cells on peripheral blood and/or bone marrow aspirate.
* Step C : Untreated patients with histologically confirmed MCL (within 3 months before baseline). The initial diagnosis has to be confirmed according to WHO classification.
* Stage II-IV in need of treatment
* ECOG performance status of 0 - 2.
* Haematology values must be within the following limits:

  1. Absolute neutrophil count (ANC)≥ 1000/mm3 independent of growth factor support
  2. Platelets ≥75,000/mm3 or ≥ 50,000/mm3 if bone marrow involvement and independent of transfusion support in either situation
* Biochemical values within the following limits:

  1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
  2. Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
  3. Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault 11) ≥ 50 mL/min/1.73m2
* HIV, anti-HBc, HbsAg test negative
* Life expectancy of more than 3 months.
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for at least 30 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer. For males, these restrictions apply for 6 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Written signed informed consent form.

Non-Inclusion criteria :

* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Major surgery within 4 weeks of inclusion.
* Known central nervous system lymphoma.
* History of stroke or intracranial haemorrhage within 6 months prior to inclusion.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
* Impaired liver, renal (GFR<50ml/min) or other organ function which will interfere with the treatment.
* Requires treatment with strong CYP3A inhibitors.
* Vaccinated with live, attenuated vaccines within 6 months of inclusion.
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. (patients HbsAg+and/or antiHBc+ and/or HIV+ are excluded)
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of study treatment (ibrutinib, GA101, GDC-0199) capsules, or put the study outcomes at undue risk.
* Known hypersensitivity to study treatment (GA101, Ibrutinib, GDC-0199) or to any of the excipients.
* Known allergy to xanthine oxidase inhibitors and rasburicase
* Severe prior reactions to monoclonal antibodies or with prior significant toxicity (other than thrombocytopenia) from Bcl-2 inhibitor
* History of prior other malignancy with the exception of: Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix at any time prior to study
* Other cancers not specified above which have been curatively treated and from which subject is disease-free for < 5 years .
* Allografted patient
* Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study.
* Pregnancy/lactation
* Men or women of reproductive potential not agreeing to use acceptable method of birth control during treatment and for 18 months after completion of treatment for the women and 6 months for the men.
* Use of any standard or experimental anti-cancer drug therapy within 28 days prior to the first dose of study drug.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Step A : occurrence of unacceptable toxicity of the combination of GA101 and Ibrutinib during the first cycle of treatment | week 4
  4 weeks after initiation of treatment.
Step B : occurrence of unacceptable toxicity (definition p3) of the combination of GA101 and Ibrutinib plus GDC-0199 during the cycle 2 in terms of Dose-Limiting Toxicities (DLTs) | At the end of cycle 2 (each cycle is 28 days)
  No unacceptable toxicity has been observed during step A, thefore the second step (step B) was initiated
Step C : occurrence of unacceptable toxicity of the combination of GA101 and Ibrutinib and GDC-0199 at the end of the cycle 2 | At the end of cycle 2 (each cycle is 28 days)
  The third step started, because no unacceptable toxicity has been observed during the second step

SECONDARY OUTCOMES:
Response (CR, PR, SD, PD) and overall response (CR+ PR) rates | 48 months
  Response (CR, PR, SD, PD) and overall response (CR+ PR) rates assessed by Cheson 99 and 07 criteria and Working Group Revised Response Criteria for Malignant Lymphomas 14
Time to progression | 48 months
Overall survival | 48 months
Safety measured by type, frequency, severity of related treatment adverse event as Assessed by CTCAE v4.0. | 48 months
Incidence of Serious Adverse Event (SAE), Adverse Event (AE) and laboratory abnormalities. | 48 months
Incidence and severity of tumor lysis syndrome | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, Pr, Principal Investigator — Nantes University Hospital
Locations (9):
- France (7):
  - CHU Angers, Angers
  - CHU de Dijon, Dijon
  - Hôpital Claude Huriez - CHRU de Lille, Lille
  - Hôpital Saint Eloi, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital du Haut Lévêque, Pessac
  - CHU Rennes, Rennes
- United Kingdom (2):
  - Derriford Hospital _ Plymouth Hospitals NHS Trust, Plymouth, Devon
  - University of Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Decombis S, Bellanger C, Le Bris Y, Madiot C, Jardine J, Santos JC, Boulet D, Dousset C, Menard A, Kervoelen C, Douillard E, Moreau P, Minvielle S, Moreau-Aubry A, Tessoulin B, Roue G, Bidere N, Le Gouill S, Pellat-Deceunynck C, Chiron D. CARD11 gain of function upregulates BCL2A1 expression and promotes resistance to targeted therapies combination in B-cell lymphoma. Blood. 2023 Nov 2;142(18):1543-1555. doi: 10.1182/blood.2023020211. PMID 37562004
- [Derived] Le Gouill S, Morschhauser F, Chiron D, Bouabdallah K, Cartron G, Casasnovas O, Bodet-Milin C, Ragot S, Bossard C, Nadal N, Herbaux C, Tessoulin B, Tchernonog E, Rossi C, McCulloch R, Gastinne T, Callanan MB, Rule S. Ibrutinib, obinutuzumab, and venetoclax in relapsed and untreated patients with mantle cell lymphoma: a phase 1/2 trial. Blood. 2021 Feb 18;137(7):877-887. doi: 10.1182/blood.2020008727. PMID 33181832